CLINICAL TRIAL: NCT06319846
Title: A Multicenter, Double-blind, Double-dummy, Randomized Clinical Trial Comparing the Efficacy and Safety of Tirofiban Versus Placebo in Preventing Recurrence of Stroke for Patients With Intracranial Artery Stenosis and High-risk Acute Non-disabling Cerebrovascular Events(CHANCE-4）
Brief Title: Tirofiban for Patients With intraCranial Artery Stenosis and High-risk Acute Non-disabling Cerebrovascular Events(CHANCE-4）
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZLRK202312
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke, Acute; TIA; Symptomatic Intracranial Artery Stenosis
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental): Initial infusion of tirofiban 0.4μg/kg body weight/minute for 30 minutes (a maximum dose of 1mg) within 24 hours of symptom onset, followed by a continuous infusion of tirofiban 0.1μg/kg body weight/minute for 48 hours.
  Interventions: Drug: Tirofiban
- Placebo group (Placebo Comparator): Initial infusion of saline placebo for 30 minutes within 24 hours of symptom onset, followed by a continuous infusion of placebo for 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirofiban — Initial infusion of tirofiban 0.4μg/kg body weight/minute for 30 minutes (a maximum dose of 1mg) within 24 hours of symptom onset, followed by a continuous infusion of tirofiban 0.1μg/kg body weight/minute for 48 hours.
  Arms: Tirofiban group
Drug: Placebo — Initial infusion of saline placebo for 30 minutes within 24 hours of symptom onset, followed by a continuous infusion of placebo for 48 hours.
  Arms: Placebo group

SUMMARY:
This is a multicenter, double-blind, double-dummy, randomized clinical trial comparing the efficacy and safety of tirofiban versus placebo in preventing recurrence of stroke for patients with intracranial artery stenosis and high-risk acute non-disabling cerebrovascular events.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, double-dummy, randomized clinical trial to assess the effects of tirofiban versus placebo in preventing recurrence of stroke at 3-month in patients with intracranial artery stenosis and high-risk acute non-disabling cerebrovascular events. The participants will receive study medication of tirofiban or placebo within 24 hours of symptom onset by a randomization ratio of 1:1. For tirofiban group - Initial infusion of tirofiban 0.4μg/kg body weight/minute for 30 minutes (a maximum dose of 1mg) within 24 hours of symptom onset, followed by a continuous infusion of tirofiban 0.1μg/kg body weight/minute for 48 hours. For placebo group - Initial infusion of saline placebo for 30 minutes within 24 hours of symptom onset, followed by a continuous infusion of placebo for 48 hours. The primary efficacy outcome is any new ischemic stroke at 3-month. The primary safety outcome is type 3 or 5 bleeding events according to the BARC criteria at 3-month.

ELIGIBILITY:
Inclusion Criteria

1. 40 years or older than 40 years;
2. Acute cerebral ischemic event due to:

   * Acute non-disabling ischemic stroke (NIHSS≤5 at the time of randomization) or,
   * TIA with moderate-to-high risk of stroke (ABCD2 score ≥ 6 at the time of randomization);
3. Accompanied with symptomatic intracranial artery stenosis, defined as ≥ 50% stenosis of the infarcted ipsilateral intracranial artery. Intracranial arteries include intracranial segments of internal carotid arteries, intracranial segments of vertebral arteries, M1-M2 segments of middle cerebral arteries, A1-A2 segments of anterior cerebral arteries, P1-P2 segments of posterior cerebral arteries, and basilar artery. The techniques for detecting intracranial artery stenosis are limited to: MRA, CTA, or DSA. The measurement for the degree of stenosis has been established by the WASID (Warfarin-Aspirin Symptomatic Intracranial Disease) study. (AJNR Am J Neuroradiol. 2000;21:643-646.);
4. Can be treated with study drug within 24 hours of symptoms onset*(*Symptom onset is defined by the "last seen normal" principle);
5. Informed consent signed.

Exclusion Criteria

1. Malformation, tumor, abscess or other major non-ischemic brain disease (e.g., multiple sclerosis) on baseline head CT or MRI.
2. Unable to complete the evaluation of intracranial artery stenosis before randomization.
3. Isolated or pure sensory symptoms (e.g., numbness), isolated visual changes, or isolated dizziness/vertigo without evidence of acute infarction on baseline head CT or MRI.
4. Iatrogenic causes (angioplasty or surgery) of minor stroke or TIA.
5. A score of > 2 on the modified Rankin scale before the symptom onset.
6. Contraindication for tirofiban:

   * Known allergy
   * Severe renal (creatinine exceeding 1.5 times of the upper limit of normal range) or hepatic (ALT or AST > twice the upper limit of normal range) insufficiency
   * Severe cardiac failure (NYHA level: III to IV)
   * History of hemostatic disorder or systemic bleeding
   * History of thrombocytopenia or neutropenia
   * History of drug-induced hematologic disorder or hepatic dysfunction
   * Low white blood cell (<2×109/L) or platelet count (<100×109/L)
7. Tirofiban has been used since this onset.
8. Hematocrit (HCT) <30%.
9. Clear indication for anticoagulation (presumed cardiac source of embolus, e.g., atrial fibrillation, prosthetic cardiac valves known or suspected endocarditis).
10. History of intracranial hemorrhage or amyloid angiopathy.
11. History of aneurysm (including intracranial aneurysm and peripheral aneurysm).
12. History of asthma or COPD (chronic obstructive pulmonary disease).
13. High-risk for bradyarrhythmia (sinus node disease, first-degree or second-degree AV block, and brady-arrhythmic syncope without pacemaker).
14. Planned or likely revascularization (any angioplasty or endovascular surgery) within the next 3 months.
15. Scheduled for surgery or interventional treatment requiring study drug cessation.
16. Severe non-cardiovascular comorbidity with life expectancy < 3 months.
17. Inability to understand and/or follow research procedures due to mental, cognitive, or emotional disorders.
18. Current treatment (last dose given within 10 days before randomization) with heparin therapy or oral anti coagulation.
19. Intravenous thrombolytic therapy (such as intravenous rtPA) or mechanical thrombectomy within 24 hours prior to randomization.
20. Participants who have large areas (greater than half of middle cerebral artery territory) of obvious low density on the baseline CT scan.
21. Gastrointestinal bleed within 3 months or major surgery within 30 days.
22. Diagnosis or suspicious diagnosis of acute coronary syndrome.
23. Participation in another clinical study with an experimental product during the last 30 days.
24. Currently receiving an experimental drug or device.
25. Pregnant, currently trying to become pregnant, or of child-bearing potential and not using birth control.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4674 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Any new ischemic stroke at 3-month | at 3-month
  Incidence of any new ischemic stroke at 3-month
Type 3 or 5 bleeding events according to the BARC criteria at 3-month | at 3-month
  Incidence of type 3 or 5 bleeding events according to the BARC criteria at 3-month

SECONDARY OUTCOMES:
Any new ischemic stroke within 1 year | within 1 year
  Incidence of any new ischemic stroke within 1 year
New clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA/ myocardial infarction/vascular death) within 3 months and 1 year; Each new vascular event will be independently evaluated. | Within 3 months after randomization and 1 year
  Incidence of new clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA/ myocardial infarction/vascular death) within 3 months and 1 year; Each new vascular event will be independently evaluated.
Disabling stroke (Modified Rankin Scale score, mRS>1) at 3 months and 1 year | at 3 months and 1 year
  Proportion of patients with disabling stroke (Modified Rankin Scale score, mRS>1) at 3 months and 1 year. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Incidence and severity of recurrent stroke and TIA | Within 3 months after randomization and 1 year
  Incidence and severity of recurrent stroke and TIA during follow-up to 3 months and 1-year (Severity is measured using a six-level ordered categorical scale that incorporates the mRS: fatal stroke/severe non-fatal stroke [mRS 4 or 5]/moderate stroke [mRS 2 or 3]/mild stroke [mRS 0 or 1]/TIA/no stroke-TIA)
Neurological impairment at 3 months (NIHSS increased≥4 from baseline ). | at 3 months
  Proportion of patients with neurological impairment at 3 months ( National Institutes of Health Stroke Scale [NIHSS] score increased≥4 from baseline).

OTHER OUTCOMES:
Type 3 or 5 bleeding events (BARC definition) at 1 year | at 1 year
  Proportion of patients with type 3 or 5 bleeding events (BARC definition) at 1 year.
Type 2, 3 or 5 bleeding events according to the BARC criteria at 3-month and 1-year. | at 3-month and 1-year
  Proportion of patients with type 2, 3 or 5 bleeding events according to the BARC criteria at 3-month and 1-year.
All bleeding events (type 1-5 bleeding events according to the BARC criteria) | at 3-month and 1-year
  All bleeding events (type 1-5 bleeding events according to the BARC criteria) at 3-month and 1-year; Each bleeding event will be independently evaluated
Total mortality at 3-month and 1-year | at 3-month and 1-year
  Proportion of patients with total mortality at 3-month and 1-year
Adverse events/Severe adverse events reported by investigators at 3-month and 1-year | at 3-month and 1-year

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - People's Hospital of Qihe County, Dezhou, Shandong
  - Liaocheng People's Hospital（Liaocheng Brain Hospital）, Liaocheng, Shandong
  - Third People's Hospital of Liaocheng, Liaocheng, Shandong
  - Yantai Penglai traditional Chinese medicine hospital, Yantai, Shandong

IPD SHARING:
Plan to Share IPD: No